CLINICAL TRIAL: NCT02425410
Title: Analysis of Viral Infections' Exposition Preceding the Type 1 Diabetes (T1D) Diagnostic in Children of the Isis-Diab Cohort. Search for Explanations of of the Disease's Early Onset
Acronym: ISIS-VIRUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre National de Génotypage (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: AOM 10061
Record Dates: First submitted 2014-08-07; First posted 2015-04-24 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus; Insulin-Dependent
Keywords: Diabetes Mellitus; Insulin-Dependent; Virus Diseases; Questionnaires; Risk assessment; Genome-Wide Association Study
MeSH Terms: conditions — Diabetes Mellitus; Virus Diseases | interventions — Genome-Wide Association Study

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood (already collected for the Isis-Diab project)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Isis-Virus: T1D patients of the Isis-Diab cohort with genetic data (GWAS) and specific environmental data on viral events during childhood
  Interventions: Other: Collect of data on viral environment of T1D patients; Genetic: Collect of blood samples for DNA extraction and genetic characterization (GWAS)

INTERVENTIONS:
Other: Collect of data on viral environment of T1D patients — Questionnaires on viral events during mother's pregnancy and patient's childhood, health book copies, addresses' geolocation, quantification of viral exposures using Sentinel Network data
Genetic: Collect of blood samples for DNA extraction and genetic characterization (GWAS) — Collect of blood samples for DNA extraction and genetic characterization (GWAS) on Illumina platform (Centre National de Genotypage)

SUMMARY:
The purpose of this study is to investigate viral factors determining the early onset of T1D. Thanks to the quantification of viral exposures of T1D patients before the disease onset with questionnaires and environmental databases analyses, and through whole genome association studies of these patients, investigators could attempt to identify gene-virus interactions determining the age of T1D onset.

DETAILED DESCRIPTION:
The "hygiene hypothesis", which has been proposed to explain the observed increase of the incidence of T1D, relies on experimental evidence acquired in mouse models. However, epidemiological data are still lacking to validate this hypothesis in man. This is critical, because -in opposition with the hygiene hypothesis- there are many reasons to believe that, at contrary, certain virus can trigger the disease.

Genetic predisposition to a severe infection form (particularly primary infection) was demonstrated for several infectious diseases (Casanova JL, Science 317:617-619, 2007; Casanova JL, EMBO J 26:915-922, 2007). It usually corresponds to deficiencies in genes involved in the host's immune response, the transmission of which being Mendelian. Genetic factors affect the ability of enteroviruses and other viruses to damage beta cells and to induce diabetes. Recently, Nejentsev et al have demonstrated a link between enteroviruses and diabetes genes: they have indeed identified 4 rare IFIH1 polymorphisms that reduce the T1D risk. However, this gene encodes an enzyme recognizing the DNA enterovirus, causing immunity activation; mutations inhibit gene activation. Except one study on HIV-1, there is to our knowledge no genome wide association studies (GWAS) in humans on the role of host's genetic polymorphisms in the risk of infection, clinical expression, duration of viral shedding, or response to therapy or to anti-viral vaccines.

We relied on our cohort of T1D children (Isis-Diab) to investigate the possible relation between viral exposures, genetic polymorphisms, and subsequent T1D.

The search for viral factors responsible for the increased T1D prevalence in youth children is difficult to implement. The absence or scarcity of infections is difficult to assess robustly at the individual level. The analysis of digestive, ENT or blood samples in the search for viruses themselves can only be done at T1D diagnosis and is therefore unlikely to be positive several years after the causal infection. It is not possible to reconstitute retrospectively viral events, which an individual has been exposed between birth and date of diabetes diagnosis. That is why our project proposes to use a proxy of viral infections crossed by a child, quantifying viral exposures to which he was submitted before the T1D diagnosis. We focused on early childhood's viral infections that may interfere with early forms of T1D. We combine 2 data sources:

* The geolocation of the child's address will locate places where he lives. Spatio-temporal data from Sentinel Network, collected since 1984, will provide access on the following viral exposures: seasonal influenza, viral diarrhea (mostly enteroviral), mumps, measles, chickenpox. If the defect of our approach is that it does not see real viral infections experienced by children, but only the level of exposure to which they were exposed according to their address, the advantage is an objective spatio-temporal description of virus epidemics around children, making it more or less likely infection of these. Only France has such Sentinel data.
* Vaccination (including MMR) and information on infectious past of children will be collected from data recorded in his book health. We will focus on the mother's pregnancy and the child between birth and 2 years of age.

Environmental data from these 2 sources will be crossed with already available genetic data from GWAS to identify gene-virus associations potentially determining age of T1D onset. This "high dimensionality" analysis will be addressed with "machine learning" programs.

If avoidable risks are identified, it would be possible to think to design clinical trials for prevention of the identified forms of T1D.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic patients included in the Isis-Diab cohort
* Patients with available genetic data (GWAS)

Exclusion Criteria:

* Patient refusal (or parents) to participate in the study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients of the Isis-Diab cohort, i.e. T1D patients aged more than 6 months, already sampled for genetic analysis.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of viral events before T1D diagnosis | From birth to 2 years
Delay between viral events and T1D diagnosis | From birth to 2 years

SECONDARY OUTCOMES:
Age at T1D diagnosis as a quantitative trait | From birth to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alain-Jacques Valleron, PhD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France; Pierre Bougnères, MD, PhD, Study Director — Inserm U986 / Pediatric endocrinology department of the Bicêtre Hospital (AP-HP)
Locations (1):
- Inserm U986, Le Kremlin-Bicêtre, France